CLINICAL TRIAL: NCT03456804
Title: An Open-Label, Parallel, Phase II Study of Single-Agent Oral ESK981 in Men With Castrate-Resistant Prostate Cancer (CRPC)
Brief Title: ESK981 in Treating Patients With Metastatic Castrate-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elisabeth Heath, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-065; NCI-2017-02330 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-065 (Other: Wayne State University/Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2018-02-09; First posted 2018-03-07 (Actual); Results first posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-06

CONDITIONS: Castration Levels of Testosterone; Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; PSA Progression; Stage IV Prostate Adenocarcinoma AJCC v7
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment ESK981 (Experimental): Patients receive pan-VEGFR/TIE2 (Vascular Endothelial Growth Factor Receptor/angopoeitin receptor2) tyrosine kinase inhibitor CEP-11981 PO QD for 5 days (Monday-Friday). Treatment repeats for up to 8 weeks in the absence of disease progression or unacceptable toxicity. If treatment is successful after 8 weeks, patients may receive up to 6 months of pan-VEGFR/TIE2 tyrosine kinase inhibitor CEP-11981.
  Interventions: Drug: ESK981

INTERVENTIONS:
Drug: ESK981 — Treatment with ESK981 for patients with metastatic castrate resistant prostate cancer

SUMMARY:
This phase II trials studies the side effects and how well ESK981 works in treating patients with castration-resistant prostate cancer that has spread to other places in the body. ESK981 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the PSA >= 50% response rate (PSA50) from baseline using the Prostate Cancer Working Group 3 (PCWG3) criteria to pan-VEGFR/TIE2 tyrosine kinase inhibitor CEP-11981 (ESK981) as a single agent in men with castration-resistant prostate cancer (CRPC) who have progressed on enzalutamide (an oral androgen-receptor inhibitor) and/or abiraterone acetate (an androgen synthesis inhibitor).

II. To assess the safety and tolerability of ESK981 as a single agent.

SECONDARY OBJECTIVES:

I. To determine the time to PSA response to ESK981 in metastatic CRPC patients. II. To determine the duration of PSA response to ESK981 in metastatic CRPC patients.

III. To determine PSA progression rates and PSA progression free survival (PFS), as defined by the PCWG3 criteria.

TERTIARY OBJECTIVES:

I. To assess exploratory biomarkers from blood and tumor biopsies.

OUTLINE:

Patients receive pan-VEGFR/TIE2 tyrosine kinase inhibitor CEP-11981 orally (PO) once daily (QD) for 5 days (Monday-Friday). Treatment repeats for up to 8 weeks in the absence of disease progression or unacceptable toxicity. If treatment is successful after 8 weeks, patients may receive up to 6 months of pan-VEGFR/TIE2 tyrosine kinase inhibitor CEP-11981.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Have signed an informed consent document indicating that the subject understands the purpose of and procedures required for the study and are willing to participate in the study
* Be willing/able to adhere to the prohibitions and restrictions specified in this protocol
* Eastern Cooperative Group (ECOG) performance status =< 1
* Patient must have evidence of castrate resistant prostate cancer as evidenced by a confirmed rising PSA (per PCWG3 criteria) and a castrate serum testosterone level (i.e. =< 50 mg/dL)
* Documented histologically confirmed adenocarcinoma of the prostate
* Metastatic prostate cancer (M1) as documented by appropriate medical imaging (i.e. computed tomography [CT]-scan, positron emission tomography [PET] scan or bone scan)
* Treatment failure of either abiraterone and/or enzalutamide as evidenced by a confirmed rising PSA (per PCWG3 criteria) and a castrate serum testosterone level (i.e. =< 50 mg/dL) while receiving treatment with either abiraterone and/or enzalutamide
* Willingness to use contraception by a method that is deemed effective by the Investigator throughout the treatment period and for at least 30 days following the last dose of therapy
* Willingness and ability to comply with study procedures and follow-up examination
* Able to swallow and retain oral medication

Exclusion Criteria:

* Current systemic therapy (other than a gonadotrophin releasing hormone [GnRH] agonist/antagonist) for CRPC including:

  * CYP-17 inhibitors (e.g. ketoconazole, abiraterone)
  * Antiandrogens (e.g. bicalutamide, nilutamide)
  * Second generation antiandrogens (e.g. enzalutamide, ARN-509, Galeterone)
  * Immunotherapy (e.g. sipuleucel-T, ipilimumab)
  * Chemotherapy (e.g. docetaxel, cabazitaxel)
* Greater than 2 lines of prior systemic therapy for CRPC
* Prior chemotherapy (e.g. docetaxel, cabazitaxel) for CRPC; prior docetaxel administered in the castrate-sensitive space is allowed
* Prior radiopharmaceutical therapy (e.g. radium-223, strontium-89, samarium-153, etc.) within the past year
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements
* Absolute neutrophil count (ANC) less than 1500/mm^3
* Platelet count less than 100000/mm^3
* Hemoglobin less than 9 g/dL
* Bilirubin greater than 1.5 times the upper limit of normal (ULN)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2.0 times the ULN in the absence of known hepatic metastases, or ALT or AST greater than 3.0 times the ULN in the presence of known hepatic metastases
* The patient has a serum creatinine value greater than 1.5 mg/dL
* The patient has active brain metastases
* The patient is currently on warfarin or heparin therapy
* The patient has any pre-existing coagulopathy, recent hemoptysis, gross hematuria, or gastrointestinal bleeding, and a history of a clinically significant cardiovascular or cerebrovascular event within 12 months prior to study entry
* The patient has uncontrolled hypertension defined as a blood pressure measurement greater than 150 mm Hg systolic or 90 mm Hg diastolic with medication
* The patient has received any investigational drug within the past 4 weeks
* The patient has previously been enrolled in the study or received ESK981
* The patient has known hypersensitivity to gelatin or lactose monohydrate
* The patient has taken a medication known to be a potent inducer of CYP1A2, CYP2C8, or CYP3A4 within 4 weeks prior to the first dose of study drug
* The patient has taken a medication known to be a potent inhibitor of CYP1A2, CYP2C8, or CYP3A4 within 2 weeks prior to the first dose of study drug

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth I. Heath, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heath EI, Chen W, Heilbrun L, Choi JE, Dobson K, Smith M, Maj T, Vaishampayan U, Kryczek I, Zou W, Chinnaiyan AM, Qiao Y. Phase II trial of multi-kinase inhibitor ESK981 in patients with metastatic castration-resistant prostate cancer. Invest New Drugs. 2024 Oct;42(5):566-574. doi: 10.1007/s10637-024-01463-x. Epub 2024 Sep 3. PMID 39227508

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment ESK981
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment ESK981
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 71 [58 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status Scale. Grade 0 to 5. 0=Normal activity, 1=Symptoms but ambulatory, 2=In bed <50% of the time, 3=In bed >50% of the time, 4=100% bedridden, 5=Dead
  Participants
    PS = 1 | 13
    PS = 0 | 0
Gleason Score [Count of Participants; unit: Participants] — Pathological scores ranging from 2 to 10, with higher numbers indicating greater risks.
  Grade 2-4 as well-differentiated tumors, Grade 5-6 as intermediately-differentiated tumors, Grade 7 as moderately to poorly differentiated tumors, Grade 8-10 as "high-grade" tumors.
  Participants
    Gleason Score 6 | 1
    Gleason Score 7 | 3
    Gleason Score 8~10 | 6
    Gleason Score unknown | 3

OUTCOME MEASURES:

1. Primary Outcome: PSA Decline of >= 50% (PSA50) From Baseline
Description: PSA decline of >= 50% (PSA50) from baseline using Prostate Cancer Working Group 3 (PCWG3) definition with point estimate and (1-sided Wilson type 90% lower) confidence interval (CI) estimates.
Time Frame: Up to 1 year
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment ESK981
Number analyzed (Participants) | 13
percentage of participants | 7.7 [1.7 to 28.2]

2. Secondary Outcome: Duration of PSA Response (RD)
Description: Will be summarized with the Kaplan-Meier (K-M) survivorship estimate. A graph of the K-M curve for RD will be generated along with the Hall-Wellner 90% confidence band, and a display of the number of patients at risk at several time points, below the X-axis. Summary statistics (6-month rate, 12-month rate, median, etc.) will be calculated from the K-M life table, each one with its respective 80% CI.
Time Frame: From start of PSA50 until PSA progression, assessed up to 1 year
Population: patients who achieved a 50% reduction in PSA from baseline
Measure: Number; unit: months
Arm/Group | Treatment ESK981
Number analyzed (Participants) | 1
months | 1.9

3. Secondary Outcome: PSA Progression Free Survival (PFS)
Description: Will be summarized with the Kaplan-Meier (K-M) survivorship estimate. A graph of the K-M curve for PFS will be generated along with the Hall-Wellner 90% confidence band, and a display of the number of patients at risk at several time points, below the X-axis. Summary statistics (6-month rate, 12-month rate, median, etc.) will be calculated from the K-M life table, each one with its respective 80% CI.
Time Frame: Date that a 25% or greater increase and an absolute increase of 2.0 ng/mL or more from the nadir is documented and confirmed by a second value obtained 3 or more weeks later, assessed up to 1 year
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment ESK981
Number analyzed (Participants) | 13
months | 0.9 [0.2 to 1.9]

4. Secondary Outcome: Time to PSA Response
Description: Will be used to summarize the time to PSA response. These descriptives will include sample size (N), median, mean, standard deviation (SD), interquartile range (IQR), minimum, and maximum.
Time Frame: From treatment start until the first documented occurrence of PSA50, assessed up to 1 year
Population: patients who achieved a 50% reduction in PSA from baseline
Measure: Number; unit: months
Arm/Group | Treatment ESK981
Number analyzed (Participants) | 1
months | 10.0

5. Other Pre Specified Outcome: Androgen Receptor (AR) Signaling
Description: Will examine the association of somatic and germline mutations with exceptional response/resistance to pan-VEGFR/TIE2 tyrosine kinase inhibitor CEP-11981.
Time Frame: Up to 1 year
Population: Measure not taken
Arm/Group | Treatment ESK981
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Circulating and Disseminated Tumor Cells as Pharmacodynamic Biomarkers
Description: Number of Circulating and disseminated tumor cells per 7.5ml as a pharmacodynamic biomarker.
Time Frame: Up to 1 year
Population: Measure not taken
Arm/Group | Treatment ESK981
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: ETS/Kinase Gene Fusions
Description: as for outcome 5
Time Frame: Up to 1 year
Population: Measure not taken
Arm/Group | Treatment ESK981
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Metastatic Kinome Activity Profiles as Predictive Biomarkers
Description: Description of immunohistochemistry of the kinases, graded 0,1,2,3
Time Frame: Up to 1 year
Population: Measure not taken
Arm/Group | Treatment ESK981
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Immunohistochemistry (IHC) of Protein Markers
Description: Ki67, Receptor, CD31, NG2, desmin, PDGFR1/2, VEGFR1/2 immunohistochemistry graded 0, 1, 2, 3
Time Frame: Up to 1 year
Population: Measure not taken
Arm/Group | Treatment ESK981
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: DNA Sequencing of Prostate Tumor
Description: copy number, Loss of heterozygosity, mutation, amplification, graded 0,1
Time Frame: Up to 1 year
Population: Measure not taken
Arm/Group | Treatment ESK981
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: An adverse event for the purposes of this protocol is the appearance of (or worsening of any pre-existing) undesirable sign, symptom, or medical condition occurring after signing the informed consent even if the event is not considered to be related to the study drug. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, related or not to the medicinal product.
Arm/Group | Treatment ESK981
All-Cause Mortality (participants affected / at risk) | 10/13
Serious Adverse Events (participants affected / at risk) | 5/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment ESK981 (N=13)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment ESK981 (N=13)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Fatigue (General disorders) | 4 (6)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (3)
General disorders and administration site condi (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Localized edema (General disorders) | 2 (2)
Lymphedema (Vascular disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Reproductive system and breast disorders - Othe (Reproductive system and breast disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT03456804/Prot_SAP_000.pdf